CLINICAL TRIAL: NCT01870440
Title: TAHOE: Sustained InTravitreal DexAmetHasone Implant (Ozurdex) for Uveitic Macular Edema
Brief Title: TAHOE: Intravitreal Dexamethasone Implant (Ozurdex) for Uveitic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern California Retina Vitreous Associates (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Rahul Khurana, M.D., Principal Investigator, Northern California Retina Vitreous Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCRVA-2013-Ozurdex-16.2
Record Dates: First submitted 2013-05-24; First posted 2013-06-06 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Macular Edema; Uveitis
Keywords: Uveitis; Macular Edema
MeSH Terms: conditions — Macular Edema; Uveitis | interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ozurdex Injection (Experimental): Ozurdex Intravitreal Injection (0.7 mg)
  Interventions: Drug: Ozurdex Intravitreal Injection (0.7 mg)

INTERVENTIONS:
Drug: Ozurdex Intravitreal Injection (0.7 mg) — Intravitreal Injection
  Other Names: Ozurdex (0.7 mg)

SUMMARY:
The purpose of this study is to determine whether an intravitreal dexamethasone implant (Ozurdex, Allergan) is effective to manage macular edema secondary to non-infectious uveitis.

DETAILED DESCRIPTION:
Uveitis accounts for more than 10% of all cases of severe vision loss in developed countries, which makes it possibly the fourth leading cause of blindness in the United States. Cystoid macular edema (CME) is the most structural complication of uveitis, resulting in visual impairment and blindness. If left untreated or undertreated over a period of years, CME may result in permanent photoreceptor damage of the macula and loss of central vision. Further, CME may persist despite adequate control of the uveitis, and therefore, adjuvant therapy to specifically treat the CME may be required.

We propose to study whether a sustained steroid delivery system (Ozurdex, Allergan) can treat uveitic macular edema. Ozurdex has been proven to be effective for non-infectious posterior uveitis; and FDA approved for posterior uveitis. The sustained delivery of the steroid and local delivery modality makes it an ideal candidate to manage macular edema in uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Uveitis CME with central subfoveal thickness > 350 microns
* non-infectious uveitis
* Visual Acuity > 20/32

Exclusion Criteria:

* Visual Acuity worse than 20/200
* Moderate or severe glaucoma (as defined as >2 topical ocular medications)
* Infectious uveitis
* Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis, vaccinia, varicella, mycobacterial infections, and fungal diseases.
* Aphakic eyes with rupture of the posterior lens capsule
* Anterior Chamber intraocular Lens and rupture of the posterior lens capsule
* Hypersensitivity to any components of the Ozurdex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (using Early Treatment Diabetic Retinopathy Study Protocal) | Day 90

SECONDARY OUTCOMES:
Central Subfoveal Retinal Thickness | Day 90
Central Subfoveal Retinal Thickness | Day 180
Best Corrected Visual Acuity | Day 180

CONTACTS AND LOCATIONS:
Locations (1):
- Northern California Retina Vitreous Associates, Mountain View, California, United States

REFERENCES:
- [Background] Lowder C, Belfort R Jr, Lightman S, Foster CS, Robinson MR, Schiffman RM, Li XY, Cui H, Whitcup SM; Ozurdex HURON Study Group. Dexamethasone intravitreal implant for noninfectious intermediate or posterior uveitis. Arch Ophthalmol. 2011 May;129(5):545-53. doi: 10.1001/archophthalmol.2010.339. Epub 2011 Jan 10. PMID 21220619